CLINICAL TRIAL: NCT04356703
Title: Impact of Prenatal Correction of Spina Bifida Using Fetoscopy and the SAFER Technique on Long-term Neurodevelopment.
Brief Title: Fetoscopic Open Spina Bifida Repair Using the SAFER Technique
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: HIAE-SAFER
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Open Spina Bifida; Myelomeningocele; Meningomyelocele; Chiari Malformation With Spina Bifida; Chiari Malformation Type 2
Keywords: myelomeningocele; spina bifida; meningomyelocele; fetal surgery; fetoscopy; fetal disease; fetal treatment
MeSH Terms: conditions — Spina Bifida Cystica; Meningomyelocele; Arnold-Chiari Malformation; Spinal Dysraphism; Fetal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children submitted to fetoscopic surgery: Children submitted to fetoscopic in utero myelomeningocele repair using the SAFER (Skin-over-biocellulose for Anternatal FEtoscopic Repair) technique will evaluate the neuropsicomotor development at 30 months of chronological age or older
  Interventions: Other: Neuropsicomotor developmental test

INTERVENTIONS:
Other: Neuropsicomotor developmental test — Children will be evaluated trough Bayley III and PEDI scale. They also will be examined by pediatrician, neurosurgeon, orthopedics and phisiatry

SUMMARY:
Children submitted to fetoscopic in utero myelomeningocele repair using the SAFER (Skin-over-biocellulose for Anternatal FEtoscopic Repair) technique will evaluate at 30 months or more, regarding ambulation, neurodevelopment, urinary and fecal status.

DETAILED DESCRIPTION:
Children submitted to fetoscopic in utero myelomeningocele repair using the SAFER (Skin-over-biocellulose for Anternatal FEtoscopic Repair) technique will evaluate the neuropsicomotor development at 30 months of chronological age. The mental evaluation will use the Bayley III and thePEDI neurodevelopmental scale. The motor development will use the difference between anatomic and motor level of the lesion. Urinary and fecal continence will be evaluated using clinical and ultrasonographic parameters. For the anatomical level determination, immaging of the spine at the lesion level will be used. Motor level and ambulation will be evaluated through standard clinical examination.

ELIGIBILITY:
Inclusion Criteria:

Children operated in utero using the SAFER technique

Exclusion Criteria:

Death before 30 month

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children submitted to prenatal repair of open spina bifida using the fetoscopic percutaneous repair technique - SAFER
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Hydrocephalus treatment - shunt or ETV | 12 months corrected age or more
  Need to treat hydrocephaly in the first year of life
Ambulation | 30 months of cronological age or more
  Ambulation Status
Neurodevelopmental test | 30 months of cronogical age or more
  PEDI scale will be performed

SECONDARY OUTCOMES:
Anatomical verus motor level | 30 months of cronological age or more
  To compare anatomical level with motor level

CONTACTS AND LOCATIONS:
Overall Officials: DENISE A LAPA, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanz Cortes M, Lapa DA, Acacio GL, Belfort M, Carreras E, Maiz N, Peiro JL, Lim FY, Miller J, Baschat A, Sepulveda G, Davila I, Gielchinsky Y, Benifla M, Stirnemann J, Ville Y, Yamamoto M, Figueroa H, Simpson L, Nicolaides KH. Proceedings of the First Annual Meeting of the International Fetoscopic Myelomeningocele Repair Consortium. Ultrasound Obstet Gynecol. 2019 Jun;53(6):855-863. doi: 10.1002/uog.20308. No abstract available. PMID 31169957
- [Background] Lapa DA. Prenatal superior to postnatal myelomeningocele surgery. J Pediatr. 2018 Jul;198:322-325. doi: 10.1016/j.jpeds.2018.04.060. No abstract available. PMID 29936963
- [Background] Lapa DA. Endoscopic fetal surgery for neural tube defects. Best Pract Res Clin Obstet Gynaecol. 2019 Jul;58:133-141. doi: 10.1016/j.bpobgyn.2019.05.001. Epub 2019 Jun 29. PMID 31350160
- [Background] Carrabba G, Macchini F, Fabietti I, Schisano L, Meccariello G, Campanella R, Bertani G, Locatelli M, Boito S, Porro GA, Gabetta L, Picciolini O, Cinnante C, Triulzi F, Ciralli F, Mosca F, Lapa DA, Leva E, Rampini P, Persico N. Minimally invasive fetal surgery for myelomeningocele: preliminary report from a single center. Neurosurg Focus. 2019 Oct 1;47(4):E12. doi: 10.3171/2019.8.FOCUS19438. PMID 31574466
- [Background] Pedreira DA, Zanon N, Nishikuni K, Moreira de Sa RA, Acacio GL, Chmait RH, Kontopoulos EV, Quintero RA. Endoscopic surgery for the antenatal treatment of myelomeningocele: the CECAM trial. Am J Obstet Gynecol. 2016 Jan;214(1):111.e1-111.e11. doi: 10.1016/j.ajog.2015.09.065. Epub 2015 Sep 18. PMID 26386383
- [Background] Herrera SR, Leme RJ, Valente PR, Caldini EG, Saldiva PH, Pedreira DA. Comparison between two surgical techniques for prenatal correction of meningomyelocele in sheep. Einstein (Sao Paulo). 2012 Oct-Dec;10(4):455-61. doi: 10.1590/s1679-45082012000400011. English, Portuguese. PMID 23386086
- [Background] Pedreira DA, Quintero RA, Acacio GL, Caldini ET, Saldiva PH. Neoskin development in the fetus with the use of a three-layer graft: an animal model for in utero closure of large skin defects. J Matern Fetal Neonatal Med. 2011 Oct;24(10):1243-8. doi: 10.3109/14767058.2011.564486. Epub 2011 Aug 17. PMID 21848412
- [Background] Sanchez e Oliveira Rde C, Valente PR, Abou-Jamra RC, Araujo A, Saldiva PH, Pedreira DA. Biosynthetic cellulose induces the formation of a neoduramater following pre-natal correction of meningomyelocele in fetal sheep. Acta Cir Bras. 2007 May-Jun;22(3):174-81. doi: 10.1590/s0102-86502007000300004. PMID 17546289